CLINICAL TRIAL: NCT07229248
Title: Drug Coated Balloon vs. Drug Eluting Stent in Young Patients With STEMI: The DCB-STEMI Randomized Trial
Brief Title: DCB vs. DES in Young STEMI Patients: The DCB-STEMI Trial
Acronym: DCB-STEMI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Professor Abdul Hakeem, Professor and Program Director, Interventional Cardiology, Director Cardiac Catheterization Labs, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NICVD IRB-32/2025
Record Dates: First submitted 2025-09-18; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: STEMI (ST Elevation MI)
Keywords: Drug coated balloon; STEMI; RCT; DES; MACE
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: Randomized, non-inferiority, parallel-group trial comparing DCB versus DES in young STEMI patients.
Who Masked: Outcomes Assessor
Masking Description: Endpoint assessment will be blinded ie the adjudication committee members will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB arm (Prevail Drug Coated Balloon) (Experimental): Patients assigned to drug coated balloon
  Interventions: Device: Drug coated balloon (Prevail; Medtronic Inc.)
- DES arm (Limus drug eluting stent) (Active Comparator): Patients receiving standard of care Drug eluting stent
  Interventions: Device: Drug eluting stent

INTERVENTIONS:
Device: Drug coated balloon (Prevail; Medtronic Inc.) — Drug coated balloon (Prevail DCB, Medtronic Inc.)
  Arms: DCB arm (Prevail Drug Coated Balloon)
Device: Drug eluting stent — standard of care
  Arms: DES arm (Limus drug eluting stent)

SUMMARY:
Background: ST Elevation Myocardial Infarction (STEMI) in young adults (<50 yrs) carries high Percutaneous coronary intervention (PCI) risks. While drug-eluting stents (DES) reduce restenosis versus angioplasty, they increase risks of in-stent restenosis, thrombosis, prolonged dual antiplatelet therapy (DAPT), and endothelial dysfunction. Drug-coated balloons (DCB) provide a "leave nothing behind" strategy, potentially mitigating these issues. Evidence, including a JACC CVI report, suggests DCB outcomes comparable to DES in STEMI. South Asia faces a heavy burden. The national Institute of Cardiovascular diseases (NICVD), Karachi performed 17,761 primary PCIs in 2022, with 45% in patients <50 yrs.

Study Design: This single-center Randomized Controlled Trial (RCT) compares paclitaxel-coated DCB (3.0 µg/mm², 30s inflation) vs. Drug eluting stents (DES) in young STEMI patients (<50 yrs) undergoing primary PCI. The primary endpoint is 1-year vessel oriented cardiac events (VOCE)= Cardiovascular /all-cause death, target vessel MI, or Target lesion revascularization (TLR). Secondary endpoints include vessel-oriented CV events, bleeding, TIMI III flow, residual stenosis, abrupt closure, and bailout stenting. An intravascular ultrasound (IVUS) substudy (100 DCB pts) will evaluate remodeling and late lumen loss (LLL) at 6 months.

Methods: 496 patients (248/arm) will be randomized 1:1, powered for non-inferiority (margin 4.5%) assuming VOCE 8.5% (DES) vs. 6.25% (DCB), 80% power, and 5% dropout. Inclusion: age 18-50, STEMI. Exclusion: End stage renal disease (ESRD), severe multivessel disease, complex lesions, or high thrombus burden. All will receive ticagrelor 90 mg BID for 1 month. A pilot of 50 pts will first assess safety (abrupt closure, lesion prep).

Analysis: Intention-to-treat (ITT) will be primary; modified ITT for secondary endpoints. Statistics include chi-square/Fisher for categorical, t-test/Wilcoxon for continuous, and Kaplan-Meier/Cox for survival. Oversight by data safety monitoring board (DSMB) and Events adjudication Committee (EAC).

Significance: This trial leverages NICVD's high PCI volume to test DCB as an alternative to DES in young STEMI patients. By avoiding permanent implants, DCB may reduce long-term complications and DAPT needs. The IVUS substudy and pilot phase strengthen rigor. If non-inferiority is proven, DCB could reshape STEMI management in South Asia and similar high-burden regions.

DETAILED DESCRIPTION:
INTRODUCTION Patients with acute myocardial infarction (AMI) are among the highest-risk patients undergoing PCI and are mostly treated with drug-eluting stents (DES). Stenting reduces elastic recoil, restenosis, and flow-limiting dissections associated with balloon angioplasty. However, it increases the risk of in-stent restenosis (ISR), bleeding from prolonged dual antiplatelet therapy (DAPT), early and late stent thrombosis, and endothelial and vasomotor dysfunction.

In young patients (<50 years), lifetime management after stenting carries unique economic and social consequences. Stent implantation means a lifelong risk of ISR, stent thrombosis, and strict adherence to DAPT-a major compliance and financial issue in this age group.

These limitations have led to the development of drug-coated balloons (DCB), which deliver antiproliferative drugs into the vessel wall without leaving a permanent implant. This "leave nothing behind" strategy is particularly attractive in young patients and those with high bleeding risk. DCBs have shown promise in ISR, small vessel disease, and STEMI. Paclitaxel-coated balloons are most commonly used, delivering 2.0-3.5 µg/mm² of paclitaxel with cytotoxicity lasting at least 14 days. With a 30-second balloon inflation, about 16% of the drug is transferred to the vessel wall, ensuring homogenous delivery while avoiding permanent implants, stent thrombosis, ISR, and prolonged DAPT.

Several studies and meta-analyses have demonstrated comparable outcomes between DCBs and DES in AMI, including STEMI. In a large multicenter analysis of STEMI patients, DCBs were associated with similar mortality and target lesion revascularization compared to DES. Other feasibility studies confirmed no excess risk of abrupt closure, thrombosis, or target vessel failure when DCBs were used in primary PCI.

Cardiovascular disease, especially AMI, remains the leading global cause of death. South Asia bears a particularly high burden, with Pakistan at the top for premature MI. The National Institute of Cardiovascular Diseases (NICVD), Karachi, has become the world's largest primary PCI center, performing 17,761 primary PCIs in 2022. Notably, 45% were in young patients (<50 years) and 12% in very young (<40 years). This provides a unique opportunity to study DCB vs DES in a high-volume RCT focused on young STEMI patients.

________________________________________ STUDY DESIGN This is a randomized controlled trial comparing DCB vs DES in young (<50 years) STEMI patients undergoing primary PCI.

Hypothesis: DCB is non-inferior to DES in reducing Vessel Oriented Composite Endpoint (VOCE) at one year.

Primary Objective: Compare 1-year VOCE between DCB and DES in young STEMI patients.

Secondary Objectives: Compare vessel-oriented CV events, target vessel failure, vessel-related MI, stent thrombosis, bleeding, TIMI III flow, residual stenosis, abrupt closure, and bailout stenting.

________________________________________ METHODS

* Design: Single-center RCT at NICVD Karachi.
* Duration: 12 months.
* Randomization: Block randomization (1:1) using sealed envelopes.
* Sample Size: 496 patients (248 per arm). Based on non-inferiority design, assuming VOCE 8.5% with DES and 6.25% with DCB, non-inferiority margin 4.5%, 80% power, 5% dropout.

Inclusion Criteria:

* Age 18-50 years
* STEMI as first coronary artery disease (CAD) presentation
* Primary PCI within 8 hours of ischemia
* Low SYNTAX score
* Killip class I-II

Exclusion Criteria:

* ESRD
* Severe 3-vessel disease or high SYNTAX score
* Complex lesions >B or large thrombus despite preparation
* Refusal of consent
* Killip III/IV
* Major bleeding history

INTERVENTIONS

* DCB Arm: Paclitaxel-coated balloon (3.0 µg/mm²), inflated for 30 seconds after adequate lesion preparation. Successful result defined as TIMI III flow, ≤30% residual stenosis, and absence of major dissection. Bailout stenting permitted if needed, but patient analyzed in DCB arm (intention-to-treat).
* DES Arm: Standard second-generation drug eluting stent with routine lesion preparation.

IVUS Substudy:

100 patients in the DCB arm will undergo IVUS at baseline, post-procedure, and 6 months to assess vessel remodeling and late lumen loss.

DAPT Protocol:

Ticagrelor 90 mg BID for 1 month post-PCI, followed by DAPT up to 1 year.

________________________________________ DATA COLLECTION & FOLLOW-UP

* Baseline demographics, risk factors, and angiographic data recorded.
* Clinical follow-up at 14 days, 30 days, 3 months, 6 months, and 12 months via visit/phone.
* Events tracked: death, MI, stent thrombosis, bleeding, stroke, repeat PCI, CABG, arrhythmias, and adverse drug reactions.
* Data captured on CRFs and stored securely.

ENDPOINTS

Primary Endpoint:

• 1-year VOCE (all-cause mortality, target vessel MI, TLR).

Secondary Endpoints:

* TIMI III flow rates
* Residual stenosis (>30% in DCB, >20% in DES)
* Bailout stenting
* Vessel-oriented events
* Bleeding

QUALITY CONTROL & ETHICS

* Ethics approval obtained from NICVD.
* Written informed consent (English/Urdu).
* Independent DSMB to monitor safety and review pilot data weekly.
* Event Adjudication Committee to validate endpoints.
* Data stored per GCP for 10 years.
* Medtronic to provide financial support but with no role in design, conduct, or analysis.

PILOT PHASE An initial pilot of 50 patients will assess safety of the DCB-only strategy in STEMI. Focus will be on lesion preparation, abrupt closure, and bailout stenting. If safe, full enrollment will proceed.

________________________________________ STATISTICAL ANALYSIS

* Population: Intention-to-treat for efficacy; modified ITT for safety.
* Categorical Variables: Chi-square or Fisher's exact.
* Continuous Variables: T-test or Wilcoxon rank-sum.
* Time-to-Event: Kaplan-Meier with log-rank test; Cox regression for hazard ratios and subgroup analysis.
* Significance: p<0.05.
* Subgroups: Age (<40 vs ≥40), sex, smoking, diabetes, renal function, weight.

SIGNIFICANCE This trial addresses a critical gap in managing young STEMI patients in South Asia, a population with extremely high disease burden and unique socioeconomic challenges. If non-inferiority of DCB is confirmed, it could reshape PCI practice by reducing long-term stent-related complications, improving compliance, and lowering financial strain in younger patients.

ELIGIBILITY:
Inclusion Criteria:

* Either gender
* Patient of age between 18 to 50 years
* Patients with STEMI ( as first presentation of CAD) undergoing Primary PCI
* Total ischemic Time less than 8 hrs.
* Low syntax score
* Stable (Killip I-II)

Exclusion Criteria:

* Patients with ESRD
* Severe 3 VD; Intermediate of High syntax score
* Lesion type>B

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 496 (Estimated)
Dates: Start 2025-11-05 (Estimated); Primary Completion 2027-12-17 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
VOCE | one year
  Composite of CV death, Target Vessel MI (including stent thrombosis) and TLR

SECONDARY OUTCOMES:
Proportion of Patients Experiencing Individual Components of Vessel-Oriented Composite Endpoint (VOCE) | one year
  The proportion of patients in each arm (DCB and DES) experiencing each individual component of VOCE (e.g., cardiac death, target vessel myocardial infarction, target lesion revascularization) will be measured at 12 months post-procedure. Events will be adjudicated by an independent clinical events committee using standardized definitions (e.g., Academic Research Consortium criteria). Data will be reported as the percentage of patients with each event in each arm, with 95% confidence intervals.
Proportion of Patients Achieving TIMI III Flow Post-Procedure | immediate post procedure
  The proportion of patients in each arm (DCB and DES) achieving Thrombolysis in Myocardial Infarction (TIMI) grade III flow (normal coronary blood flow) immediately post-procedure will be assessed via coronary angiography using standardized angiographic criteria. Data will be reported as the percentage of patients with TIMI III flow in each arm, with 95% confidence intervals
Proportion of Patients with Angiographic Residual Stenosis Exceeding Thresholds (>30% for DCB, >20% for DES) | Immediate post procedure
  The proportion of patients with residual stenosis (percentage of vessel diameter narrowing) exceeding 30% in the DCB arm and 20% in the DES arm will be measured via coronary angiography immediately post-procedure. Data will be reported as the percentage of patients exceeding the respective thresholds in each arm, with 95% confidence intervals.
Rate of Abrupt Vessel Closure Post-Procedure | within 24 hours post procedure
  The rate of abrupt vessel closure (complete occlusion of the target vessel) in each arm (DCB and DES) will be assessed via coronary angiography during the index procedure or within 24 hours post-procedure. Closure events will be confirmed by the event adjudication committee. Data will be reported as the percentage of patients experiencing abrupt vessel closure in each arm, with 95% confidence intervals.
Proportion of Patients Requiring Bail-Out Stenting in the DCB Arm | intra procedure
  The proportion of patients in the DCB arm requiring bail-out stenting due to inadequate procedural results (e.g., residual stenosis >50%, dissection, or abrupt closure) during the index procedure will be recorded. Bail-out stenting will be determined by the treating physician and verified by procedural reports. Data will be reported as the percentage of patients in the DCB arm requiring bail-out stenting, with 95% confidence intervals.
Proportion of Patients with BARC Type 3, or 5 Bleeding Events | 12 months
  The proportion of patients in each arm (DCB and DES) experiencing Bleeding Academic Research Consortium (BARC) type 3 (overt bleeding with hemoglobin drop or requiring intervention), or type 5 (fatal bleeding) events will be assessed at [12 months] post-procedure. Bleeding events will be adjudicated by an independent clinical events committee using BARC criteria. Data will be reported as the percentage of patients with BARC 3, or 5 bleeding in each arm, with 95% confidence intervals.

OTHER OUTCOMES:
Mean Late Lumen Loss in the DCB Arm at 6 Months Post-Procedure | 6 months
  We seek to evaluate 100 randomized patients of the DCB arm to establish baseline IVUS features prior to DCB after DCB at the completion of the procedure and at 6 months follow up.
  Primary IVUS Outcome (for the substudy) Late lumen loss (LLL) will be calculated as the difference between the minimum lumen diameter (MLD, in millimeters) measured by intravascular ultrasound (IVUS) immediately post-procedure and the MLD at 6-month follow-up in the DCB arm. IVUS will be performed using a standardized protocol by an independent core laboratory. LLL will be reported as the mean ± standard deviation (SD) across the 100 randomized patients in the DCB arm, with 95% confidence intervals.
Mean Minimum Lumen Diameter in the DCB Arm at Baseline, Post-Procedure, and 6 Months | Baseline (pre-DCB), immediately post-procedure, and 6 months post-procedure
  Minimum lumen diameter (MLD) will be measured by intravascular ultrasound (IVUS) at three time points: baseline (pre-DCB), immediately post-procedure, and at 6-month follow-up in the DCB arm. IVUS measurements will be conducted by an independent team using standardized software. MLD will be reported as the mean ± standard deviation (SD) for each time point across the 100 randomized patients in the DCB arm, with 95% confidence intervals. Changes in MLD between time points will be analyzed using paired t-tests or equivalent non-parametric tests.
Mean Percent Diameter Stenosis in the DCB Arm at Baseline, Post-Procedure, and 6 Months | Baseline (pre-DCB), immediately post-procedure, and 6 months post-procedure
  Percent diameter stenosis (%DS) will be calculated by intravascular ultrasound (IVUS) as (reference vessel diameter- minimal lumen diameter/ reference vessel diameter x 100) at three time points: baseline (pre-DCB), immediately post-procedure, and at 6-month follow-up in the DCB arm. IVUS measurements will be performed by an independent team using standardized software. %DS will be reported as the mean ± standard deviation (SD) for each time point across the 100 randomized patients in the DCB arm, with 95% confidence intervals. Changes in %DS between time points will be analyzed using paired t-tests or equivalent non-parametric tests.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Hakeem, MD, Principal Investigator — NICVD
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request and submission to the PI. The proposition will be formally reviewed by the steering committee.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication of the results untill 2 hours.
Access Criteria: IPD will be shared upon reasonable request and submission to the PI. The proposition will be formally reviewed by the steering committee.

REFERENCES:
- [Result] Mangner N, Farah A, Ohlow MA, Mobius-Winkler S, Weilenmann D, Wohrle J, Linke A, Stachel G, Markovic S, Leibundgut G, Rickenbacher P, Cattaneo M, Gilgen N, Kaiser C, Scheller B, Jeger RV; BASKET-SMALL 2 Investigators. Safety and Efficacy of Drug-Coated Balloons Versus Drug-Eluting Stents in Acute Coronary Syndromes: A Prespecified Analysis of BASKET-SMALL 2. Circ Cardiovasc Interv. 2022 Feb;15(2):e011325. doi: 10.1161/CIRCINTERVENTIONS.121.011325. Epub 2022 Jan 10. PMID 35000455
- [Result] Huang KN, Grandi SM, Filion KB, Eisenberg MJ. Late and very late stent thrombosis in patients with second-generation drug-eluting stents. Can J Cardiol. 2013 Nov;29(11):1488-94. doi: 10.1016/j.cjca.2013.04.001. Epub 2013 Jul 4. PMID 23830291
- [Result] McKavanagh P, Zawadowski G, Ahmed N, Kutryk M. The evolution of coronary stents. Expert Rev Cardiovasc Ther. 2018 Mar;16(3):219-228. doi: 10.1080/14779072.2018.1435274. Epub 2018 Feb 5. PMID 29381087